CLINICAL TRIAL: NCT03682679
Title: Use Sonoelastography to Predict the Reparability of Large-to-massive Rotator Cuff Tears
Brief Title: Sonoelastography to Predict Rotator Cuff Tears
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CMRPG8H0811
Record Dates: First submitted 2018-09-18; First posted 2018-09-25 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2020-02

CONDITIONS: Rotator Cuff Tear
Keywords: large-to-massive rotator cuff tears; reparability; sonoelastography; magnetic resonance imaging
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Sonoelastography — This diagnostic test would be executed by a physician who has experiences of using Siemens Acuson S2000 ultrasound system for more than three year. The examination includes two of four rotator cuff muscles, listed as follows, supraspinatus muscle and infraspinatus muscle. Linear transducer (4-9 MHz) would be used for the whole test. The probe would be positioned along the longitudinal axis of the muscle belly. Compressive sonoelastography technique is used for semiquantitative analysis. In order to maintain the quality of images, quality factor needs to be over or equal to 60. The quantitative analysis was performed by shear wave sonoelastography and the region of interest (ROI) would be divided into four quadrants. The physicians will measure the shear wave velocity at the center point of each quadrant.

SUMMARY:
Large-to-massive rotator cuff tears accounts for 30% of all rotator cuff tears. These problems can be solved by surgeries, but only part of them can be completely repaired. The prognosis for partial repair is worse than complete repair, so evaluating the possibility of complete repair is so important that it will affect the decision of treatment. More and more recent researches focused on using magnetic resonance imaging (MRI) for evaluation of fatty infiltration of rotator cuff muscles to predict the reparability of large-to-massive rotator cuff tears. However, the availability of MRI is not that good as ultrasound, so some researchers are starting to use ultrasound to predict the reparability of large-to-massive rotator cuff tears. Because it is hard to observe the tissue quality through the general ultrasound, many researchers use sonoelastography to evaluate the tissue elasticity and viability. This aim of this study is to:

1. check the reliability of sonoelastography.
2. associate the findings of sonoelastography to the results of MRI.
3. build a predictive model for the reparability of large-to-massive rotator cuff tears.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are diagnosed with rotator cuff tear by an orthopedist.
2. The large-to-massive rotator cuff tears need to be confirmed by magnetic resonance imaging or ultrasound. The definitions of this diagnosis include a tear over 3 cm or any full-thickness of tears in more than two rotator cuff muscles.
3. Being willing to cooperated with the arranged examinations before the operation.

Exclusion Criteria:

1. Patients who are only diagnosed with partial-thickness rotator cuff muscle tears or small- to large- sized full-thickness tears.
2. Patients who have acromioclavicular arthritis that needs distal clavicle resection.
3. Patients who had serious glenohumeral arthritis, pseudoparalysis, or any other shoulder trauma history.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigator will enroll participants with diagnosis of large-to-massive rotator cuff tears who will receive surgical repairs later, and sonoelastography and MRI are necessary for preoperative evaluation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Sonoelastography | Baseline
  This diagnostic test would be executed by a physician who has experiences of using Siemens Acuson S2000 ultrasound system for more than three year. The examination includes two of four rotator cuff muscles, listed as follows, supraspinatus muscle and infraspinatus muscle. Linear transducer (4-9 MHz) would be used for the whole test. The probe would be positioned along the longitudinal axis of the muscle belly.
  Compressive sonoelastography technique is used for semiquantitative analysis. In order to maintain the quality of images, quality factor needs to be over or equal to 60. The quantitative analysis was performed by shear wave sonoelastography. While assessing, the region of interest (ROI) would be divided into four quadrants. The physicians will measure the shear wave velocity for wight times at the center point of each quadrant.

SECONDARY OUTCOMES:
Passive range of motions | Baseline
  Passive range of motions of internal and external rotation, abduction, extension, and flexion, which are assessed by a goniometer.
Muscle strength | Baseline
  Muscle strength assessment include the following motions, which are internal and external rotation, abduction, extension, and flexion. They are measured by a manual dynamometer.
American Shoulder and Elbow Surgeons score. | Baseline
  Shoulder function that are scaled by using American Shoulder and Elbow Surgeons score.
MRI | Baseline
  MRI was performed on a 1.5T system (Signa Horizon LX, GE Healthcare) equipped with a standard shoulder surface coil. The shoulder MRI protocol was identical for all patients and consisted of axial proton-density-weighted fast spin-echo with fat suppression sequence, the sequences was performed above the level o f the acromioclavicular joint down to below the axillary pouch with the following parameters: Coronal oblique proton-density-weighted with and without fat suppression, with axis parallel to the supraspinatus tendon, and sagittal oblique proton-density--weighted with and without fat suppression, with axis perpendicular to the coronal oblique axis, the ast spin-echo sequences were performed with the following parameters: TR msec/TE msec, 2700-4800 /25-40, echo-train length, 6; matrix, 256 × 256; field of view, 180 mm; section thickness, 2.5 mm with 2-mm gap. No IV or intraarticular gadolinium was administered.
Surgical outcome | Baseline
  The investigator will discuss the surgical outcome with the orthopedist to define whether the tear side is repaired partially or completely. If the tendon can be repaired using simple side-to-side tendon repair, horizontal mattress transosseous repair via the bone trough and reduced into an anatomic position, or via the rough area of greater tuberosity (marginal converging repair), it is defined as complete repair of the tendon. If the tendon cannot be reduced to the anatomic footprint and the orthopedist only secures re-attachment of the infraspinatus to the posterior side of greater tuberosity and/or the subscapularis of lesser tuberosity, it is defined as partial repair of the tendon.
B-mode ultrasound | Baseline
  The ultrasound machine will be calibrated similarly using the musculoskeletal (MSK) preset and B-mode with autogain. The dynamic range will be set at 70 dB for all participants. The examiners will apply adequate transducer pressure to obtain optimal images for comparisons of muscle and bone echo. The Heckmatt scale will be used to grade the muscle echogenicity within each ROI of supraspinatus and infraspinatus muscles. The grading rule is as follows:
  1. Grade 1: Normal
  2. Grade 2: Increased muscle echo intensity with distinct bone echo
  3. Grade 3: Marked increased muscle echo with reduced bone echo
  4. Grade 4: Very strong muscle echo and complete loss of bone echo

CONTACTS AND LOCATIONS:
Overall Officials: Po-Cheng Chen, MD, Study Chair — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Tseng YH, Chou WY, Wu KT, Chang CD, Chen YC, Huang YC, Lin WC, Chen PC. Use sonoelastography to predict the reparability of large-to-massive rotator cuff tears. Medicine (Baltimore). 2020 Jul 2;99(27):e21139. doi: 10.1097/MD.0000000000021139. PMID 32629749